CLINICAL TRIAL: NCT04021030
Title: Building Collaborations to Address Drug Problems in the United States and China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Medicine - PKUHSC Joint Institute for Translational and Clinical Research (Unknown); Peking University (Other); Meridian Health Services (Unknown)
Responsible Party: Principal Investigator, Mark A. Ilgen, Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00122412
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (CBT) (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The therapeutic intervention consists of 8, one-hour individual therapy sessions delivered over the course of 2 to 4 weeks with a trained CBT therapist. These sessions are designed to provide beneficial coping strategies that are helpful in dealing with both chronic pain and substance use.

SUMMARY:
The purpose of this study is to evaluate the impact of a Cognitive Behavioral Therapy (CBT) intervention on the distribution and variability of pain level before and after intervention receipt among people with co-occurring chronic pain and Substance Use Disorders (SUDs) over a three-month follow-up period.

DETAILED DESCRIPTION:
The project is an open trial of the CBT intervention for 20 adults receiving detoxification treatment with comorbid pain. Participants will be screened for pain and other conditions by completing a self-report survey questionnaire. Eligible participants will be asked to complete a baseline assessment. A trained research therapist will conduct individual therapy with participants twice a week for 2-4 weeks. Participants will be re-assessed at 1- and 3-month post-intervention follow-ups to track changes in their pain, functioning, and substance use.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Currently receiving detoxification treatment
* Report pain of at least moderate or greater intensity over the three months prior to baseline assessment as indicated by an average score of four or greater on the Numeric Rating Scale (NRS)
* Have access to a phone for confidential personal therapy after the completion of detoxification treatment. For individuals who enter the residential treatment at the facility following the detoxification treatment, a research therapist will meet with them in person at a private office at the facility during their stay due to program's restriction on phone usage.

Exclusion Criteria:

* Inability to speak and understand English
* Inability to give informed, voluntary, written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with decrease in pain level ≥ 18 % (or two points) on the Numeric Rating Scale (NRS) | 3 months post-intervention
  Pain level will be assessed using the Numeric Rating Scale (NRS). The NRS is a 0-10 scale, with higher scores indicating greater intensity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ilgen, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Meridian Health Services, Waterford, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentiﬁcation (text, tables, ﬁgures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Data access requests should be directed to Mark Ilgen (PI) at marki@umich.edu up to 36 months following article publication. To gain access, requestors will be required to sign a Data Access Agreement.